CLINICAL TRIAL: NCT07167875
Title: Personalized Digital Behavior Change Interventions to Optimize Oral Hygiene Behaviors: Randomized Controlled Trial
Brief Title: Personalized Digital Coaching for Oral Hygiene Adherence: Randomized Controlled Trial.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Vivek Shetty, DDS, DMD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-24-0661; UH3DE028723 (NIH)
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dental Disease; Behavioral Changes
Keywords: dental disease; digital interventions; behavioral changes
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention (Experimental): Participants randomized to the intervention group will receive a personalized digital coaching promoting adherence to the 2x2x4 brushing routine.
  Interventions: Behavioral: Personalized Digital Oral Health Coaching
- traditional oral hygiene instruction (No Intervention): All participants will use an electronic toothbrush and mobile app to record brushing behavior throughout the study. However, the control arm will use the devices strictly for data collection without access to personalized digital coaching features.

INTERVENTIONS:
Behavioral: Personalized Digital Oral Health Coaching — All participants will use an electronic toothbrush and mobile app to record brushing behavior throughout the study. However, only the intervention arm will receive personalized digital coaching through the Oralytics app, including tailored feedback, educational messages, and motivational prompts.
  Arms: Digital Intervention

SUMMARY:
The goal of this clinical trial is to learn if a personalized Digital Oral Health Intervention (DOHI) improves how well adults follow recommended tooth brushing routines. Researchers also aim to understand which factors influence the success of the intervention.

The main questions this study will answer are:

Does using the DOHI lead participants to brush twice daily for two minutes, covering all four quadrants (the 2x2x4 routine) more consistently than traditional oral hygiene instructions alone?

Which participant characteristics, such as demographics or baseline oral hygiene habits, affect how well the DOHI helps people improve their brushing?

How does engagement with the digital coaching and technology impact adherence to recommended oral hygiene practices?

In this study:

230 adults receiving care at community dental clinics in California will participate.

Everyone will begin with a 2-week run-in period using traditional oral care instructions.

Afterward, participants will be randomly assigned to one of two groups:

The control group will continue with traditional oral hygiene instructions.

The intervention group will receive traditional oral hygiene instructions plus personalized digital coaching delivered through a mobile app and an electronic toothbrush system.

The DOHI provides personalized feedback, educational content, and motivational prompts that adapt over time based on each participant's brushing behavior and engagement.

Both groups will use an electronic toothbrush to objectively record when, how long, and how well they brush.

Participants will:

Follow the assigned oral hygiene instructions for 19 weeks.

Use an electronic toothbrush and mobile app as instructed.

Have their brushing data automatically collected and analyzed by researchers.

The study will look at changes in brushing frequency and duration from before to after the intervention. Researchers will also explore how personal characteristics and engagement with technology influence outcomes.

The results of this trial will help community dental clinics know if personalized, digital coaching can help more adults maintain healthy habits and achieve better oral health, and guide future improvements in digital health interventions for oral hygiene.

DETAILED DESCRIPTION:
This multisite randomized controlled trial is designed to evaluate whether a personalized Digital Oral Health Intervention (DOHI) can improve adherence to recommended oral hygiene behaviors compared to traditional oral hygiene instruction alone. The study addresses the persistent challenge of maintaining long-term oral hygiene habits by utilizing technology-facilitated coaching, adaptive intervention delivery, and reinforcement learning algorithms that respond to each participant's real-time brushing behaviors.

A total of 230 adults (aged 18 years and older) will be recruited from three community dental clinics in California: Dientes Community Dental Care (Santa Cruz County), Petaluma Health Center (Sonoma County), and University of California, Los Angeles (UCLA)Dental Clinics (Los Angeles County). Following baseline education in the recommended 2x2x4 brushing protocol (brushing twice daily for two minutes, covering all four dental quadrants) and a 2-week run-in period to ensure comfort with the electronic toothbrush system and study procedures, eligible participants will be randomized in equal numbers to either the intervention or control group.

Participants in the control group will continue with traditional oral hygiene instruction and receive standard feedback on their brushing patterns over the 19-week intervention period. The intervention group will also receive traditional instruction and standard feedback, but in addition they will be provided with personalized digital coaching through the DOHI platform. The DOHI integrates an electronic toothbrush and the Oralytics mobile application to deliver tailored feedback, educational resources, and motivational strategies such as micro-incentives. The system uses reinforcement learning algorithms to dynamically adjust the timing, frequency, and content of coaching prompts based on each participant's brushing data and engagement patterns, aiming to optimize involvement and support sustainable behavior change.

The primary outcome of the study is the change in participants' adherence to the recommended brushing frequency and duration, objectively measured from baseline through 19 weeks using data collected by the electronic toothbrush system. Secondary outcomes include analyses of individual-level factors-such as demographics, initial oral hygiene behaviors, and patterns of technology use-that may influence the effectiveness of the DOHI for promoting oral self-care.

The results of this trial are expected to provide evidence for the implementation of adaptive digital interventions to support oral health, with the potential for broad application in community dental care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Fluent in English (speaking, reading, writing)
* Dentulous or partially edentulous (minimum 2 teeth per quadrant)
* Own and regularly use a smartphone (iOS or Android) with active data plan
* Receiving dental care at a participating study site
* Willing to use electronic toothbrush and mobile application for 19 weeks
* Able to provide informed consent

Exclusion Criteria:

* Edentulous (no natural teeth)
* Fewer than 18 teeth or fewer than 2 teeth in any quadrant
* Unable to use mobile devices due to cognitive or physical impairments
* Unwilling to comply with study procedures
* Current participation in another oral health intervention study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Brushing Sessions as Measured by Electric Toothbrush Data Collection | 19 weeks
  Change in number of daily brushing sessions from baseline to 19 weeks, objectively measured through electric toothbrush data collection system. Baseline defined as average daily brushing frequency during 2-week run-in period. Target adherence is twice daily brushing (2 sessions per day).
Mean Change in Daily Brushing Duration as Measured by Electric Toothbrush Data Collection | 19 weeks
  Change in average brushing duration per session measured in minutes from baseline to 19 weeks using electric toothbrush data collection. Baseline defined as mean brushing duration during 2-week run-in period. Target duration is 2 minutes per session. Data reported as mean change in minutes with standard deviation.

SECONDARY OUTCOMES:
Demographic Predictors of Digital Oral Health Intervention Response as Measured by Multivariable Logistic Regression Analysis | 19 weeks
  Analysis of demographic factors (age, gender, race/ethnicity, education level, income, employment status) that predict differential response to the Digital Oral Health Intervention (DOHI) compared to control group using multivariable logistic regression models. Response defined as binary outcome: achieving ≥75% adherence to recommended 2x2x4 brushing routine (success) versus <75% adherence (failure) measured by electronic toothbrush data collection over 19 weeks. Analysis will examine interaction effects between demographic variables and treatment assignment. Results reported as odds ratios with 95% confidence intervals for each demographic predictor, indicating the strength of association between specific demographic characteristics and likelihood of intervention success. Higher odds ratios indicate greater likelihood of achieving target adherence for participants with that demographic characteristic.
Baseline Oral Hygiene Behavior Predictors of Digital Intervention Success as Measured by Electronic Toothbrush Data Collection and Multivariable Regression Analysis | 19 weeks
  Investigation of baseline oral hygiene behaviors that predict successful adherence to the Digital Oral Health Intervention (DOHI) using multivariable regression analysis. Baseline predictors include: brushing frequency (sessions per day), brushing duration (minutes per session), timing patterns (morning/evening consistency), and oral health knowledge scores assessed via validated questionnaire during 2-week run-in period. Success defined as composite binary outcome: achieving both ≥1 additional brushing session per day AND ≥30 seconds increase in average brushing duration from baseline to 19 weeks, measured objectively by electronic toothbrush data collection system.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Shetty, DMD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Petaluma Health Center-Dental, Petaluma, CA, Petaluma, California
  - Dientes Community Dental Care, Santa Cruz, California

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available to the research community 12 months after publication of primary analyses. External data requests require written proposals and institutional oversight documentation, subject to confidentiality agreements and Principal Investigator approval.
Time Frame: Data will be available beginning 12 months after publication of primary results and ending 5 years after article publication
Access Criteria: Requests for data access require written scientific proposals, institutional oversight documentation, and signed data use agreements. Requests will be reviewed by the Principal Investigator and institutional data sharing committee."